CLINICAL TRIAL: NCT06493708
Title: Effectiveness of Eye Movement Desensitization and Reprocessing (EMDR) Applied to Borderline Personality Disorder: a Randomized-controlled Single-blind Study in a Real-world Care Setting
Brief Title: Effectiveness of EMDR in Borderline Personality Disorder: a RCT Single-blind Study in a Real-world Care Setting
Acronym: EMBODIER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Antonio Vita, Prof, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: EMDR2023-02
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR intervention (Experimental): 14 sessions of psychotherapy with EMDR will be carried out with patients. One session per week, lasting 90 minutes. The first two sessions will be used for the description of the EMDR method and for stabilization, then there will be treatment sessions.
  Interventions: Other: Trauma focused psychotherapy: EMDR
- Waiting List (No Intervention): Treatment as usual

INTERVENTIONS:
Other: Trauma focused psychotherapy: EMDR — 14 sessions of psychotherapy with EMDR will be carried out with patients. One session per week, lasting 90 minutes. The first two sessions will be used for the description of the EMDR method and for stabilization, then there will be treatment sessions.
  Arms: EMDR intervention

SUMMARY:
Borderline personality disorder (BPD) is a severe mental disorder characterized by four major symptomatological domains: interpersonal instability, perceptive and identity disorders, emotional and behavioural dysregulation. Considering a multifactorial etiological model, it has been suggested that the interaction between behavioral, environmental and genetic factors may promote the development of BPD. Early life stress events (ELS) in childhood and adolescence are highly prevalent in this population and constitute an environmental risk factor for the development of BPD. This correlates with the fact that Post-traumatic Stress Disorder (PTSD) is frequently comorbid in BPD leading to more severe symptoms and worse psychosocial functioning. At the therapeutic level, the treatment of BPD is an open challenge as psychotherapeutic interventions are of limited effectiveness and characterized by high drop-out rates. Eye Movement Desensitization and Reprocessing (EMDR) is the gold standard for treating PTSD. However, scientific evidence on the application of EMDR in patients with BPD is limited. This study aims to assess the feasibility and effectiveness of an EMDR protocol on the nuclear symptomatology of BPD (emotional and behavioral dysregulation) in a group of DBP patients with/without PTSD comorbidity, through a systematic assessment of the peculiar dimensions of the disorder. The basic hypothesis is that EMDR, through a short-term intervention, can act both on the traumatic PTSD-like experiences reported by patients and on the clinical manifestations peculiar to DBP, in particular by improving the emotional regulation capacity of patients with BPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be over 18 years old
* A current diagnosis of PBD according to the DSM-5 was confirmed using the SCID-5-CV and SCID-5-PD diagnostic scale

Exclusion Criteria:

* Suicidal ideation in the last 3 months (suicidal thoughts active intentionally but without specific planning or suicidal thoughts active with planning and intentionality)
* Intellectual disability
* Any active disturbance from use of substances or alcohol
* Any other diagnosis of Axis I, except for Depressive Disorders, Anxious Spectrum Disorders, Obsessive-Compulsive Disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Core symptoms of BPD | 4 timepoints: baseline (T0), after 6 (T6), 12 (T12), 18 (T18) weeks
  The primary outcome is the improvement of the core symptoms of BPD, measured by the Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD)

SECONDARY OUTCOMES:
Self perception of BPD symptoms | 4 timepoints: baseline (T0), after 6 (T6), 12 (T12), 18 (T18) weeks
  Self perception of BPD symptoms measured by the Borderline Symptom List 23 (BSL-23).

OTHER OUTCOMES:
Emotion disregulation | 4 timepoints: baseline (T0), after 6 (T6), 12 (T12), 18 (T18) weeks
  Emotion disregulation measured by the Difficulties in emotion regulation scale (DERS-36)
Ruminative thinking | 4 timepoints: baseline (T0), after 6 (T6), 12 (T12), 18 (T18) weeks
  Ruminative thinking measured by the Rumination Response Scale (RRS)
Dissociative symptoms | 4 timepoints: baseline (T0), after 6 (T6), 12 (T12), 18 (T18) weeks
  Dissociative symptoms measured by the Dissociative Experiences Scale (DES)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Minelli, Prof, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- ASST Spedali Civili Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes